CLINICAL TRIAL: NCT05594342
Title: Effects of Adding Ivabradine in Patients With Cardiogenic Shock Requiring Inotropic Support
Brief Title: Ivabradine Effects in Cardiogenic Shock Requiring Inotropic Support
Acronym: IVA-CS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Young Investigator Group of Cardiovascular Research (Network)
Responsible Party: Principal Investigator, Abdallah Almaghraby, Associate Professor of Cardiology, The Young Investigator Group of Cardiovascular Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YIG-10202201
Record Dates: First submitted 2022-10-04; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure; Cardiogenic Shock; Ischemic Heart Disease
Keywords: Heart Failure; Cardiogenic shock; Ivabradine
MeSH Terms: conditions — Heart Failure; Shock, Cardiogenic; Myocardial Ischemia | interventions — Ivabradine; Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivabradine+ dobutamine infusion (Experimental): Patients will receive ivabradine 7.5 mg twice daily via oral route after starting dobutamine infusion by 30 minutes.
  Interventions: Drug: Ivabradine 7.5Mg Tab; Drug: DOBUTamine Injectable Solution
- Dobutamine infusion only (Active Comparator): Patient will receive dobutamine infusion only for cardiogenic shock
  Interventions: Drug: DOBUTamine Injectable Solution

INTERVENTIONS:
Drug: Ivabradine 7.5Mg Tab — Patients will receive ivabradine 7.5 mg twice daily via oral route after dobutamine infusion by 30 minutes.
  Other Names: Ivabradine
  Arms: Ivabradine+ dobutamine infusion
Drug: DOBUTamine Injectable Solution — Dobutamine infusion by a dose that is titrated according to blood pressure Ranging from 5 to 20 ug/kg/minute
  Other Names: Dobutamine

SUMMARY:
Data regarding the safety and efficacy of ivabradine use in severely decompensated HFrEF requiring inotropic support is limited to case series.1 This study aimed to evaluate ivabradine safety and tolerability in admitted cardiogenic shock patients who started on dobutamine infusion for inotropic support.

DETAILED DESCRIPTION:
Background and study rationale:

Ivabradine is a Heart Rate (HR) lowering agent which acts by inhibiting the If current in the sinoatrial node. It is currently indicated in patients with chronic heart failure with reduced ejection fraction (HFrEF). Dobutamine is an inotropic drug used in cardiogenic shock patients and it is associated with an increase in HR and incidence of cardiac arrhythmias.2 However, studies have suggested that increased heart rate may be deleterious in decompensated HFrEF due to an inverted Bowditch-Treppe response. Data regarding the safety and efficacy of ivabradine use in severely decompensated HFrEF requiring inotropic support is limited to case series.1, 2

Aim of the work:

* This study aims to evaluate ivabradine safety and tolerability in admitted cardiogenic shock patients who started on dobutamine infusion for inotropic support.
* Design: Randomized open-label interventional clinical trial.

Methods and patients:

* Study Type: Interventional (Clinical Trial)
* Estimated Enrollment: 200 participants
* Allocation: Randomized
* Perspective: Prospective Study
* Intervention Model: Two Group Assignment
* Masking: None (Open Label)
* Primary purpose: Treatment
* Official title: Ivabradine effects in cardiogenic shock requiring inotropic support (IVA-CS)
* Start Date: 01 August 2022
* Estimated Primary Completion Date: 01 January 2023

ELIGIBILITY:
Inclusion Criteria:

* Decompensated heart failure with reduced ejection fraction (HFrEF) admitted for cardiogenic shock requiring inotropic support.

Exclusion Criteria:

* Decompensated heart failure with reduced ejection fraction (HFrEF) not requiring inotropic support.
* Patients with no oral intake
* Patients who refused to sign the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Heart rate reduction | Up to 7 days
  Amount of reduction of heart rate calculated by subtracting the heart rate at the time of weaning from the initial heart rate
Time of weaning from dobutamine infusion | Up to 7 days
  The time needed to completely wean dobutamine infusion calculated in hours
Duration of hospital stay | Up to 1 month
  Total duration of hospital stay calculated in days

SECONDARY OUTCOMES:
Ventricular arrhythmias (Ventricular Tachycardia and/or Fibrillation) | Up to 1 month
  Any ventricular arrhythmias will be documented
Supraventricular arrhythmia | Up to 1 month
  Any supraventricular arrhythmias will be documented

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Andalusia Hospitals, Alexandria
  - Tiba Hospital, Alexandria

IPD SHARING:
Plan to Share IPD: Undecided